CLINICAL TRIAL: NCT06697041
Title: Clinical and Laboratory Factors for the Progression of Severe Dengue Among Hospitalized Patients During an Upsurge
Acronym: PROSED
Status: Completed | Type: Observational
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: PR-23077
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Dengue Fever With Warning Signs
Keywords: dengue; severe dengue; warning sign; plasma leakage; dengue hemorrhagic fever
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — CBC will be carried out in the CLS hematology lab by a Sysmex hematology analyzer as per the SOP approved by the accredited authority. The clinical Hematology Lab will perform the reference NS1 dengue antigen and IgM-IgG antibody RDT as per their SOP.
  Molecular serotyping will be conducted at IDD's Emerging Infections & Parasitology Laboratory. The CDC DENV-1-4 RT-PCR Assay, an in-vitro diagnostic platform, has received approval from the US Food and Drug Administration (FDA) for identifying dengue in individuals exhibiting mild or severe dengue symptoms. The test's primers and probes have been meticulously designed to detect presently circulating strains of DENV-1-4 with a sensitivity comparable to strains found globally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis (if any): Not applicable Objectives: To identify factors for progression to severe Dengue in hospitalized patients.

Methods: Prospective Observational study

DETAILED DESCRIPTION:
Global perspective:

Mosquito-borne dengue is a global public health issue in the tropics and subtropics. Dengue is endemic in over 100 countries, according to WHO. Around 40% of the world's population-3.6 billion-lives in dengue-endemic areas. Dengue infects 400 million people, sickens 100 million, and kills 21,000 each year. In studies of acute febrile illness in US visitors returning from South-central and Southeast Asia, South America, Mexico, and the Caribbean, dengue is the main cause due to increased international travel and the popularity of dengue-endemic destinations. Thus, dengue-related US hospitalizations are rising. Prevention methods, such as early detection and prompt clinical therapy, can lower case fatality rates from 10% to <1%.

National perspective:

Dengue has been hyperendemic in Bangladesh since 2000. The current dengue spike is exceptional in its seasonality and an early fast increase compared to past years, which began in late June. According to WHO, this year's case fatality rate is 0.47%, higher than usual. However, Bangladeshi clinical spectrum, serotype predominance, novel and modified serotypes (DEVN-5), and immunological responses need more research. However, future dengue prevention and treatment techniques require serotype-specific clinical and laboratory indicators and immune reactivity in distinct spectrums.

This research is conducted in hospitals to identify the burden of severe dengue and its link to dengue fever in our country. Dengue fever is now managed supportively without antiviral medication. The cause of severe and potentially deadly dengue is unknown. Prior DENV exposure, co-morbidity, and genetic predisposition may increase the risk of severe dengue sickness. The study results will help us understand and solve the problem. The aim is to assess the clinical and laboratory parameters related to severe Dengue and the transition from non-severe to severe Dengue in hospitalized Bangladeshis.

Primary objectives: To identify factors for progression to severe Dengue in hospitalized patients.

Secondary objectives:

1. To determine the circulating dengue serotype (DENV-1, DENV-2, DENV-3, DNEV-4, and others) about different spectrums of dengue fever in Bangladesh.
2. To determine primary and secondary immune responses (IgG and IgM) following dengue infection [by examining IgG to IgM ratio (ELISA) with analyzing of DENV NS1 IgG subclass types (ELISA)] and the association of immune responses to the different spectrum of dengue fever in Bangladesh.
3. To characterize specific laboratory biomarkers (hematocrit level, white blood cell count, platelet count, coagulation profile, serum albumin level, liver enzymes, LDH) and immunological parameters (NS1, IgM, and IgG) associated with severe Dengue cases.
4. Verbal autopsy and retrospective analyses of death cases from the respective hospital.
5. To explore physicians' barriers and challenges in treating Dengue and identify and develop the best treatment approaches through formative research.

Study design: Observational Cohort study Study sites: Four sites/hospitals: Dhaka North City Corporation Hospital (DNCCH), Mugda Medical College and Hospital (MuMCH), Dhaka Medical College Hospital (DMCH), and Dhaka Hospital of icddr,b.

Study population: >1 year Study period: The study lasts from 1 January 2024 to 31 June 2024. Total enrolment will be for 6 months or until the estimated patient enrolment is fulfilled.

Study Activities:

Screening: The study nurse and health worker will identify eligible patients during hospital admission. After meeting enrolment requirements, the caregiver or attendance will be asked for informed written consent. After consenting, the patient will be enrolled. Patients will give a full history, and the study nurse will record it in CRF. Socio-demographic, household, co-morbidity, and medical history will be recorded.

Clinical monitoring and recording: The study physician will record four hourly vital signs and warning signals in the case report form. Nurses and the study site night physician will record vitals during the night shift trial. Warning indicators will be operationally defined. The project research physician will do a tourniquet test during enrollment. An axillary temperature of 38°C or above indicates fever.

Laboratory investigations: DMCH, MuMCH, and DNCC blood samples will be delivered to icddr,b laboratory for reference value consistency. DMCH, MuMCH, and DNCC admitting physicians will receive the results via WhatsApp group on the same day and receive paper copies for patient files.

Blood samples will be taken from research participants at enrollment, discharge, or deterioration and on day 21 (18-28 days) during recovery. If fever is present on day 5 or 6, 2.5 ml of blood will be drawn for IgM and IgG. Diarrhea patients included will also provide stool samples. The IEDCR and icddr,b labs will be tested. Under-5s can collect 10 ml of blood, while adults can collect 15 ml. Within 6 hours of collection, serum tests should be refrigerated at -70°C. The hospital policy requires sterile plastic tubes to collect l specimens from diarrheal patients at Dhaka Hospital.

A qualitative assessment of experienced healthcare professionals from selected hospitals will examine their real-life experiences with treatment (including symptom management, hospitalization, and recovery), treatment options (including traditional medicines, alternative therapies, and other local remedies), challenges/barriers to treatment, gaps in current treatment approaches, and patient and health care professional preferences. One Research Officer (RO) with an Anthropology degree and qualitative research experience will choose participants and conduct interviews under the supervision of a senior Anthropologist. RO will choose qualitative interviewees based on their dengue treatment experience at the specified hospitals and variety. Eight Key Informant Interviews (KII) will be conducted with dengue treatment professionals from four hospitals. In addition, in-depth interviews (IDIs) will be conducted with eight physicians and eight nurses actively treating at the selected hospitals to understand current treatment practices and best treatment approaches to replicate elsewhere to improve treatment, especially for vulnerable populations. After data saturation, the number of interviews will be calculated.

A verbal autopsy will be performed on every death if the caregiver consents. Then, the study personnel will retrospectively evaluate death instances, collect data, and arrange verbal autopsy from caregivers at DNCC hospital.

Calculating Sample Size: This study's sample size was calculated in two steps to reach a 5% progression of severe dengue. This calculation ensures that the study has the statistical power to identify the effect size and whether clinical and laboratory parameters affect severe Dengue development. First, a minimum sample size of 321 was calculated. Thus, if 321 patients are included, 16 (5% of 321) will have severe Dengue cases, and 305 will be non-severe.

Data analysis: Data management and statistical analyses will use STATA (16.0) and SPSS for Windows. The dataset will be summarized using frequency (%), mean, standard deviation, median, and interquartile range. Statistical plots will be employed to illustrate data distribution and identify outliers. When appropriate, chi-squared or Fisher's Exact tests compare categorical variables, whereas Mann-Whitney tests compare continuous variables.

Multivariable logistic regression will examine the relationship between binary outcomes (e.g., severe Dengue vs. non-severe Dengue) and predictor factors (e.g., age, sex, admission sickness status, laboratory test findings). To measure association strength, odds ratios (OR) and 95% confidence intervals (CI) will be calculated. Statistical significance is evaluated at p-value < 0.05.

Thematically analyzing verbal autopsy data will reveal dengue-related death trends. Formative study data will be thematically coded to understand treatment approaches and their feasibility. Post-study beginning, a formal Statistical Analysis Plan (SAP) will guide the analysis process, providing openness and rigor.

The expedited committee of the Research Review Committee (RRC) and Ethical Review Committee (ERC) of icddr,b will review the study protocol, data collection tools, and informed consent forms before starting the study. The study will follow the 'Declaration of Helsinki' (2000), ICH, Tripartite Guidelines, and GCP. These protocols protect the rights and integrity of study participants, conduct all study procedures correctly, collect enough data, document it, and verify it.

No patient benefit is expected beyond routine therapy and monitoring. The study only poses a modest risk to participants during blood collection. No additional specimens will be taken for this investigation. Bengali will be used to write and structure the permission form for study subjects without formal education. The patient and study subject's accompanying person will hear the consent form if they cannot read it. The participant can leave the research and decline to answer any questions. This hospital will treat the patient as usual if they refuse the research. Patient data will be kept private, anonymous, and secret. Our study staff will have exclusive access to all medical information, treatment descriptions, and laboratory test results from the specific ward.

Labs accredited for testing:

The International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b) employs multidisciplinary international and national scientists. It has adequate facilities to treat shock, severe sepsis, and electrolyte abnormalities caused by diarrhea. Dhaka Hospital of icddr,b contains an intensive care section for critically unwell children. A 24-hour backup generator, refrigerator (-20°C), and deep freezer (-80°C) are available. All study-related research can be done at the biochemistry laboratory, which is open 24/7.

ELIGIBILITY:
Inclusion Criteria:

* Dengue fever with warning signs with Ns1 positive and or IgM positive
* Informed written consent or assent.

Exclusion Criteria:

* Severe dengue during screening or denied consenting

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will enroll adults > over 18 from all four study sites. In addition, children from 1 year to 17 years old will be enrolled at Dhaka North City Corporation Hospital. Any patients complaining of fever between 2-6 days with features suggestive of dengue, such as severe headache, retro-orbital pain, myalgia, arthralgia, transient macular or maculopapular rash, minor hemorrhagic manifestations, (petechiae, ecchymosis, purpura, epistaxis, bleeding gums, haematuria, or a positive tourniquet test), facial flushing or erythema, injected oropharynx, anorexia
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Host factors & comorbidities | January 01- June 30; 2025
  Association with age, sex, co-morbid condition, care seeking behaviours
Laboratory infection markers and immune parameters | 01/01/2024 to 30/06/2025
  Laboratory biomarkers, immune factor, serotyping
Sociodemographic factors | On admission
  Resident, occupation, monthly income, living condition, health-seeking behaviors
Clinical progression parameters during hospitalization | January 01, 2024 to December 31, 2024
  Clinical sign symptoms during admission and then differences at final outcome, such as on discharge or in death.

CONTACTS AND LOCATIONS:
Overall Officials: Lubaba Shahrin, MBBS, FCPS, Principal Investigator — Scientist, ICDDRB
Locations (1):
- International Centre for Diarrheal Disease Research Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
The participants identifiers will be anonymous at all the stages of the research

REFERENCES:
- [Background] Wang SM, Sekaran SD. Early diagnosis of Dengue infection using a commercial Dengue Duo rapid test kit for the detection of NS1, IGM, and IGG. Am J Trop Med Hyg. 2010 Sep;83(3):690-5. doi: 10.4269/ajtmh.2010.10-0117. PMID 20810840
- [Background] Guzman MG, Alvarez M, Halstead SB. Secondary infection as a risk factor for dengue hemorrhagic fever/dengue shock syndrome: an historical perspective and role of antibody-dependent enhancement of infection. Arch Virol. 2013 Jul;158(7):1445-59. doi: 10.1007/s00705-013-1645-3. Epub 2013 Mar 8. PMID 23471635
- [Background] Mustafa MS, Rasotgi V, Jain S, Gupta V. Discovery of fifth serotype of dengue virus (DENV-5): A new public health dilemma in dengue control. Med J Armed Forces India. 2015 Jan;71(1):67-70. doi: 10.1016/j.mjafi.2014.09.011. Epub 2014 Nov 24. PMID 25609867
- [Background] Changal KH, Raina AH, Raina A, Raina M, Bashir R, Latief M, Mir T, Changal QH. Differentiating secondary from primary dengue using IgG to IgM ratio in early dengue: an observational hospital based clinico-serological study from North India. BMC Infect Dis. 2016 Nov 28;16(1):715. doi: 10.1186/s12879-016-2053-6. PMID 27894268
- [Background] Vicente CR, Herbinger KH, Froschl G, Malta Romano C, de Souza Areias Cabidelle A, Cerutti Junior C. Serotype influences on dengue severity: a cross-sectional study on 485 confirmed dengue cases in Vitoria, Brazil. BMC Infect Dis. 2016 Jul 8;16:320. doi: 10.1186/s12879-016-1668-y. PMID 27393011
- [Background] Delli Ponti R, Mutwil M. Structural landscape of the complete genomes of dengue virus serotypes and other viral hemorrhagic fevers. BMC Genomics. 2021 May 17;22(1):352. doi: 10.1186/s12864-021-07638-7. PMID 34000991
- [Background] Tsheten T, Clements ACA, Gray DJ, Adhikary RK, Furuya-Kanamori L, Wangdi K. Clinical predictors of severe dengue: a systematic review and meta-analysis. Infect Dis Poverty. 2021 Oct 9;10(1):123. doi: 10.1186/s40249-021-00908-2. PMID 34627388
- [Background] Ng WY, Atan R, Mohd Yunos N, Bin Md Kamal AH, Roslan MH, Quah KY, Teh KX, Zaid M, Kassim M, Mariapun J, Ngim CF, Dhanoa A, Yeo TW. A double whammy: The association between comorbidities and severe dengue among adult patients-A matched case-control study. PLoS One. 2022 Sep 20;17(9):e0273071. doi: 10.1371/journal.pone.0273071. eCollection 2022. PMID 36126060
- See also: International Centre for Diarrheal Disease Research Bangladesh — https://www.icddrb.org
- Available data/document: Anonymous dataset upor request by scientific use. Data will be shared by the Institutional Review Board.: Lubaba Shahrin — https://www.icddrb.org — https://www.icddrb.org